CLINICAL TRIAL: NCT04598711
Title: Effects of Remote Limb Ischemic Conditioning to Enhance Muscle Power, Dynamic Balance, and Walking Performance in Children With Cerebral Palsy
Brief Title: Ischemic Conditioning to Enhance Function (I-C-FUN) in Children With Cerebral Palsy
Acronym: I-C-FUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Swati Manoharrao Surkar, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-003232
Record Dates: First submitted 2020-10-01; First posted 2020-10-22 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are masked to group assignment (RLIC vs. Sham conditioning) and the assessor will be masked to group assignment of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote Limb Ischemic Conditioning (RLIC) (Experimental): RLIC is achieved via blood pressure cuff inflation to at least 20 mmHg above systolic blood pressure to 200 mmHg on the more involved thigh. RLIC involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. RLIC is performed on visits 1-14.
  Interventions:
  * Behavioral: RLIC
  * Behavioral: Muscle power training
  * Behavioral: Balance training
  * Behavioral: Treadmill training
  Interventions: Behavioral: RLIC; Behavioral: Muscle Power training; Behavioral: Balance training; Behavioral: Treadmill Training
- Sham Conditioning (Sham Comparator): Sham conditioning is achieved via blood pressure cuff inflation to 25 mmHg on the more involved thigh. Sham involves 5 cycles of 5 minutes blood pressure cuff inflation followed by alternating 5 minutes of cuff deflation and requires 45 minutes. Sham conditioning is performed on visits 1-14.
  Interventions:
  * Behavioral: RLIC
  * Behavioral: Muscle power training
  * Behavioral: Balance training
  * Behavioral: Treadmill training
  Interventions: Behavioral: Sham Conditioning; Behavioral: Muscle Power training; Behavioral: Balance training; Behavioral: Treadmill Training

INTERVENTIONS:
Behavioral: RLIC — See descriptions under arm/group descriptions. RLIC is delivered for 14 visits. Visits 1-3 occur on consecutive work days and visits 4-14 occur on alternating week days.
  Other Names: Remote Limb Ischemic Conditioning
  Arms: Remote Limb Ischemic Conditioning (RLIC)
Behavioral: Sham Conditioning — See descriptions under arm/group descriptions. Sham conditioning is delivered for 14 visits. Visits 1-3 occur on consecutive work days and visits 4-14 occur on alternating week days.
  Other Names: Sham
  Arms: Sham Conditioning
Behavioral: Muscle Power training — All participants undergo power training of the quadriceps muscles using unilateral and bilateral leg presses (Total Gym GTS, San Diego, CA), 3 times/week for 4 consecutive weeks (12 sessions). Power training will follow standard American College of Sports Medicine guidelines for frequency, intensity, progression etc. Power training is provided at visits 3-14.
  Other Names: Quadriceps power training
Behavioral: Balance training — All participants undergo training on a balance board, learning to hold the board level with equal weight on each leg. Participants perform the balance task for 15, 30-second trials per day at visits 3-14.
  Other Names: Dynamic Stability Platform Training
Behavioral: Treadmill Training — All participants will undergo short burst interval treadmill training using self-selected and fast walking speeds.
  Other Names: Gait training

SUMMARY:
The purpose of this research study is to determine if remote limb ischemic conditioning (RLIC) can increase skeletal muscle power, enhance learning of motor (dynamic balance) task, and improve walking performance in children with cerebral palsy (CP).

DETAILED DESCRIPTION:
Ischemic conditioning is a phenomenon in which an organ exposed to a controlled, short-term, local, sublethal ischemia protects from subsequent ischemia. Remote ischemic conditioning is another more practical approach where transient ischemia and reperfusion applied to a remote organ or tissue, protects other organs or tissues from further episodes of lethal ischemia/reperfusion injury. Remote limb ischemic conditioning (RLIC) is a clinically feasible way of performing remote ischemic conditioning where alternating, brief ischemia and reperfusion is delivered with cyclic inflation and deflation of a blood pressure cuff on the arm or leg.

The overall goal of this research is to use ischemic conditioning to enhance muscle power, motor leaning, and mobility in children with CP. Our previous work demonstrated that when paired with strength training, RLIC improved muscle strength and activation in healthy, young adults and motor learning in healthy older adults. The current study extends that work to determine if RLIC enhances muscle power, dynamic balance, and walking performance in children with CP. This Phase II study will yield the necessary information to design and execute subsequent randomized controlled trials in children with CP as well as other neurological conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with unilateral or diplegia cerebral palsy (CP)
2. Gross Motor Function Classification System (GMFCS) levels I-III

Exclusion Criteria:

1. Children with other developmental disabilities such as autism, developmental coordination disorders, etc.
2. Children with cognitive deficits or communication problem
3. Children with balance disorders such as vestibular disorders, posterior fossa tumors etc.
4. Children with known cardiorespiratory dysfunctions
5. Children who are receiving other adjunct therapies such as TMS, tDCS, vagal nerve stimulation
6. Presence of lower extremity condition, injury, or surgery which could compromise conditioning and training
7. Children with sickle cell disease

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Peak knee extension power | Pre-intervention to 1 month post-intervention follow-up
  Power is defined as the ability to exert a maximum force in short amount of time (speed) while performing knee extension. Bilateral quadriceps power will be measured using Humac Norm Isokinetic testing device (Computer Sports Medicine Inc, Stoughton, MA).
Change in Balance Score | Pre-intervention to 1 month post-intervention follow-up
  The average amount of time in seconds that a participant maintains the stability platform within ±5° of horizontal position during 15 trials of 30 seconds each. The total score will range between 0-30 seconds. Higher balance score indicates better balance performance.
Change in Walking Speed | Pre-intervention to 1 month post-intervention follow-up
  Self-selected and fast walking speeds will be measured using 10-meter walk test.

SECONDARY OUTCOMES:
Quadriceps Electromyography | Pre-intervention to 1 month post-intervention follow-up
  While performing the isokinetic power testing, the electromyography (EMG) data will be recorded simultaneously. The EMG data will be used to quantify the electrical amplitude of quadriceps muscle.
Gait Analysis | Pre-intervention to 1 month post-intervention follow-up
  Lower extremity walking kinematics and kinetics will be measured using 10-camera motion analysis system (Qualisys Inc., Gothenburg, Sweden). Specific kinematic variables are hip, knee, and ankle joint torques. Kinetic variables are peak hip, knee, and ankle sagittal plane joint moments.
Lower limb activity | Pre-intervention to 1 month post-intervention follow-up
  Lower extremity activity will be measured using accelerometers (Actigraphs) worn on bilateral ankles for 24 hours. Specific accelerometry variable will be number of steps.

CONTACTS AND LOCATIONS:
Overall Officials: Swati M Surkar, PT, PhD, Principal Investigator — Assistant Professor, East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
After completion of the study, all of the individual participant data after de-identification will be submitted to East Carolina University data repository.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available soon after the completion of the study.
Access Criteria: Contact Dr. Surkar

REFERENCES:
- [Background] Gidday JM. Cerebral preconditioning and ischaemic tolerance. Nat Rev Neurosci. 2006 Jun;7(6):437-48. doi: 10.1038/nrn1927. PMID 16715053
- [Background] Saxena P, Newman MA, Shehatha JS, Redington AN, Konstantinov IE. Remote ischemic conditioning: evolution of the concept, mechanisms, and clinical application. J Card Surg. 2010 Jan-Feb;25(1):127-34. doi: 10.1111/j.1540-8191.2009.00820.x. Epub 2009 Jun 22. PMID 19549044
- [Background] Kharbanda RK, Nielsen TT, Redington AN. Translation of remote ischaemic preconditioning into clinical practice. Lancet. 2009 Oct 31;374(9700):1557-65. doi: 10.1016/S0140-6736(09)61421-5. PMID 19880021
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Meng R, Asmaro K, Meng L, Liu Y, Ma C, Xi C, Li G, Ren C, Luo Y, Ling F, Jia J, Hua Y, Wang X, Ding Y, Lo EH, Ji X. Upper limb ischemic preconditioning prevents recurrent stroke in intracranial arterial stenosis. Neurology. 2012 Oct 30;79(18):1853-61. doi: 10.1212/WNL.0b013e318271f76a. Epub 2012 Oct 3. PMID 23035060
- [Background] Ali ZA, Callaghan CJ, Lim E, Ali AA, Nouraei SA, Akthar AM, Boyle JR, Varty K, Kharbanda RK, Dutka DP, Gaunt ME. Remote ischemic preconditioning reduces myocardial and renal injury after elective abdominal aortic aneurysm repair: a randomized controlled trial. Circulation. 2007 Sep 11;116(11 Suppl):I98-105. doi: 10.1161/circulationaha.106.679167. PMID 17846333
- [Background] Liu ZJ, Chen C, Li XR, Ran YY, Xu T, Zhang Y, Geng XK, Zhang Y, Du HS, Leak RK, Ji XM, Hu XM. Remote Ischemic Preconditioning-Mediated Neuroprotection against Stroke is Associated with Significant Alterations in Peripheral Immune Responses. CNS Neurosci Ther. 2016 Jan;22(1):43-52. doi: 10.1111/cns.12448. Epub 2015 Sep 19. PMID 26384716
- [Background] Jean-St-Michel E, Manlhiot C, Li J, Tropak M, Michelsen MM, Schmidt MR, McCrindle BW, Wells GD, Redington AN. Remote preconditioning improves maximal performance in highly trained athletes. Med Sci Sports Exerc. 2011 Jul;43(7):1280-6. doi: 10.1249/MSS.0b013e318206845d. PMID 21131871
- [Background] Kjeld T, Rasmussen MR, Jattu T, Nielsen HB, Secher NH. Ischemic preconditioning of one forearm enhances static and dynamic apnea. Med Sci Sports Exerc. 2014 Jan;46(1):151-5. doi: 10.1249/MSS.0b013e3182a4090a. PMID 23846166
- [Background] de Groot PC, Thijssen DH, Sanchez M, Ellenkamp R, Hopman MT. Ischemic preconditioning improves maximal performance in humans. Eur J Appl Physiol. 2010 Jan;108(1):141-6. doi: 10.1007/s00421-009-1195-2. Epub 2009 Sep 18. PMID 19760432
- [Background] Bailey TG, Jones H, Gregson W, Atkinson G, Cable NT, Thijssen DH. Effect of ischemic preconditioning on lactate accumulation and running performance. Med Sci Sports Exerc. 2012 Nov;44(11):2084-9. doi: 10.1249/MSS.0b013e318262cb17. PMID 22843115
- [Background] Surkar SM, Bland MD, Mattlage AE, Chen L, Gidday JM, Lee JM, Hershey T, Lang CE. Effects of remote limb ischemic conditioning on muscle strength in healthy young adults: A randomized controlled trial. PLoS One. 2020 Feb 4;15(2):e0227263. doi: 10.1371/journal.pone.0227263. eCollection 2020. PMID 32017777
- [Background] Sutter EN, Mattlage AE, Bland MD, Cherry-Allen KM, Harrison E, Surkar SM, Gidday JM, Chen L, Hershey T, Lee JM, Lang CE. Remote Limb Ischemic Conditioning and Motor Learning: Evaluation of Factors Influencing Response in Older Adults. Transl Stroke Res. 2019 Aug;10(4):362-371. doi: 10.1007/s12975-018-0653-8. Epub 2018 Aug 7. PMID 30088217
- [Background] Damiano DL, Laws E, Carmines DV, Abel MF. Relationship of spasticity to knee angular velocity and motion during gait in cerebral palsy. Gait Posture. 2006 Jan;23(1):1-8. doi: 10.1016/j.gaitpost.2004.10.007. Epub 2005 Jan 7. PMID 16311188
- [Background] Steele KM, Damiano DL, Eek MN, Unger M, Delp SL. Characteristics associated with improved knee extension after strength training for individuals with cerebral palsy and crouch gait. J Pediatr Rehabil Med. 2012;5(2):99-106. doi: 10.3233/PRM-2012-0201. PMID 22699100
- [Background] Steele KM, van der Krogt MM, Schwartz MH, Delp SL. How much muscle strength is required to walk in a crouch gait? J Biomech. 2012 Oct 11;45(15):2564-9. doi: 10.1016/j.jbiomech.2012.07.028. Epub 2012 Sep 5. PMID 22959837
- [Background] Moreau NG, Holthaus K, Marlow N. Differential adaptations of muscle architecture to high-velocity versus traditional strength training in cerebral palsy. Neurorehabil Neural Repair. 2013 May;27(4):325-34. doi: 10.1177/1545968312469834. Epub 2013 Jan 4. PMID 23292847
- [Background] Hyngstrom AS, Murphy SA, Nguyen J, Schmit BD, Negro F, Gutterman DD, Durand MJ. Ischemic conditioning increases strength and volitional activation of paretic muscle in chronic stroke: a pilot study. J Appl Physiol (1985). 2018 May 1;124(5):1140-1147. doi: 10.1152/japplphysiol.01072.2017. Epub 2018 Feb 8. PMID 29420152
- [Background] Cherry-Allen KM, Gidday JM, Lee JM, Hershey T, Lang CE. Remote limb ischemic conditioning enhances motor learning in healthy humans. J Neurophysiol. 2015 Jun 1;113(10):3708-19. doi: 10.1152/jn.01028.2014. Epub 2015 Apr 1. PMID 25867743
- [Background] Christie A, Kamen G. Short-term training adaptations in maximal motor unit firing rates and afterhyperpolarization duration. Muscle Nerve. 2010 May;41(5):651-60. doi: 10.1002/mus.21539. PMID 19941348

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04598711/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT04598711/ICF_001.pdf